CLINICAL TRIAL: NCT06582004
Title: Comparisons of the Effects and Clinical Outcomes of CH2 Vaginal Gel Versus Placebo on CIN1 With High-risk HPV Patients: A Prospective Randomized Controlled Trial
Brief Title: Comparisons of the Effects and Clinical Outcomes of CH2 Vaginal Gel Versus Placebo on CIN1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202405043RSD
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Cervical Intraepithelial Neoplasia; Human Papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): use vaginal hyaluronic acid gel as placebo
  Interventions: Dietary Supplement: Placebo hyaluronic acid gel
- CH2 vaginal gel (Experimental): use CH2 vaginal gel as intervention The usage frequency is 2 units per week, with a 3-day interval between each unit, for a total duration of 24 weeks
  Interventions: Dietary Supplement: CH2 vaginal gel

INTERVENTIONS:
Dietary Supplement: CH2 vaginal gel — The usage frequency is 2 units per week, with a 3-day interval between each unit, for a total duration of 24 weeks
  Arms: CH2 vaginal gel
Dietary Supplement: Placebo hyaluronic acid gel — The usage frequency is 2 units per week, with a 3-day interval between each unit, for a total duration of 24 weeks
  Arms: Placebo

SUMMARY:
In Taiwan, Pap smear screen has been offered every year for women over 30 years old since 1995. The incidence of cervical invasive cancer decreased from 25/100,000 person in 1995 to 7.0/100,1000 person in 2016. In contrast, the incidence of pre-cancerous lesions increased gradually. According to ASCCP, observation and repeated cytology in 6-12 months is recommended in colposcopy-diagnosed CIN1 patients. Most of the low-grade lesions regressed spontaneously without treatment; 49 percent of CIN1 regressed to negative in six months, and 70 percent regressed in 12 months.

Emerging evidence suggests associations between the composition of the vaginal microbiota (VMB), human papillomavirus (HPV) infection, and cervical intraepithelial neoplasia (CIN). Previous research included 87 patients with untreated CIN2. It reported that patients with a Lactobacillus-dominant microbiome at baseline are more likely to have regressive disease at 12 months. Lactobacillus spp. depletion and presence of specific anaerobic taxa are associated with CIN2 persistence and slower regression. 82.9 percent of women with low-grade squamous intraepithelial lesions (LSIL) tested positive for HPV. CH2 vaginal gel is a marketed health product derived from natural ingredients, including water, probiotic glycerol, and plant extracts. Investigators have designed this trial to compare the following outcomes between participants who use and those who use placebo: 1. the regression rate of CIN1, 2. the time to regression of CIN1, and 3. the HPV clearance rate in participants.

DETAILED DESCRIPTION:
Emerging evidence suggests associations between the composition of the vaginal microbiota (VMB), human papillomavirus (HPV) infection, and cervical intraepithelial neoplasia (CIN). 82.9% of women with CIN1 tested positive for HPV. CH2 vaginal gel is a marketed health product derived from natural ingredients, including water, probiotic glycerol, and plant extracts. The hypothesis is that this product will improve the vaginal environment and microbiota, leading to increased HPV clearance, and enhancing the regression rate of CIN1. Investigators have designed this trial to compare outcomes between participants who use CH2 and those who use placebo.

Patients and Methods:

Investigators will conduct a prospective randomized controlled study to enroll 50 participants with CIN1 from the Gynecologic colposcopy clinic of National Taiwan University Hospital. Participants will be randomly assigned to receive either CH2 vaginal gel or none. All enrolled patients will be assessed before use, at three months post-use, and at six months post-use, including questionnaire surveys, ThinPrep Pap tests, and HPV genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals aged 20 years (inclusive) or older who have abnormal Pap smear results and have been diagnosed with CIN1 via colposcopy biopsy, and are also positive for high-risk HPV. This includes:
* Patients with Pap smear results of CIN2, ASCUS, or CIN1 who have undergone colposcopic biopsy of suspicious lesions or random biopsies, with pathology confirming CIN1.
* Patients with Pap smear results of CIN1 who have undergone colposcopic biopsy of suspicious lesions or random biopsies, and where the biopsy sample is insufficient for diagnosis or the biopsy pathology is normal.

Exclusion Criteria:

* Female patients who are currently pregnant, planning to become pregnant, or are underage.
* Patients with an allergy to the ingredients in CH2 Natural Purifying Protection Serum.
* Patients diagnosed with CIN2, CIN3, or higher through colposcopic biopsy.
* Patients with urinary tract or pelvic infections.
* Patients with significantly impaired cognitive function.
* Patients who are unable to self-administer vaginal gel.
* Patients with immunocompromised conditions, end-stage liver or kidney disease, those using steroids, or those who have previously undergone total hysterectomy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
pap smear result | up to 9 months
  Thinprep smear every 3 months. The report from thinprep smear and coloposcope examination. Data will be categorized as CIN1, CIN2 and above, inflammation, normal.

SECONDARY OUTCOMES:
HPV clearance rate | up to 9 months
  Cervical swab for high risk HPV test

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hau Chen, Principal Investigator — National Taiwan University Hospsital
Locations (1):
- National Taiwan University Hospital, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No